CLINICAL TRIAL: NCT01125579
Title: NEURAPAS Balance in Children With Nervous Restlessness, e.g. Agitated Depression
Brief Title: Effectiveness of NEURAPAS Balance in Children With Nervous Restlessness
Status: Completed | Type: Observational
Sponsor: Pascoe Pharmazeutische Praeparate GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 162A07NPB
Record Dates: First submitted 2010-05-14; First posted 2010-05-18 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2010-05

CONDITIONS: Nervousness; Restlessness; Depression (Agitated); Affective Disorders
Keywords: nervousness; restlessness; depression; affective disorder
MeSH Terms: conditions — Psychomotor Agitation; Depression; Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children aged 6-12: Children suffering from nervous restlessness, e.g. in agitated depression (ICD 10, F3 and DSM IV "affective disorders"), aged 6-12 years

SUMMARY:
Purpose: To document data on effectiveness of NEURAPAS® balance (NPB) in the treatment of nervous restlessness in children aged 6 to 12.

Each patient is treated with NPB. No placebo group is established. Course and severity of symptoms is documented by a questionnaire on 13 common symptoms of nervous restlessness and a Visual Analogue Scale (VAS). A standardized questionnaire (Parent Child Behaviour Checklist (CBCL/4-18)) is completed. Choice and doses of therapy are at the respective physician's discretion. The planned treatment and observation period is 2 - 4 weeks.

DETAILED DESCRIPTION:
Purpose: To document data on effectiveness of NEURAPAS® balance (NPB) in the treatment of nervous restlessness in children aged 6 to 12.

Patients and methods: A prospective, non-interventional, non-randomized, observational study conducted in German pediatric practices. Each patient is treated with NPB. No placebo group is established. As subjective criteria to document course and severity of symptoms, a questionnaire on 13 common symptoms of nervous restlessness and a Visual Analogue Scale (VAS) is used. As an objective criterion, a standardized questionnaire (Parent Child Behaviour Checklist (CBCL/4-18)) is completed. Choice and doses of therapy are at the respective physician's discretion. The planned treatment and observation period is 2 - 4 weeks.

ELIGIBILITY:
Due to the design as an Observational Study no inclusion or exclusion criteria are named. The included patient group is described under "Cohort / Group".

Observational Criteria:

* age 6 - 11 (extremes included)
* nervous restlessness and/or
* agitated depression and/or
* affective disorders

Exclusion Criteria:

* patients <6 and >12 years of age

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 6 - 11 (extremes included) suffering from nervous restlessness and/or agitated depression according to ICD-10 F3 and DSM-IV "affective disorders"
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2008-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Change in Parent Child Behaviour Checklist (CBCL/4-18) | after 2 + 4 weeks´ treatment
  Parent Child Behaviour Checklist (CBCL/4-18), standardized questionnaire

SECONDARY OUTCOMES:
Tolerability of NEURAPAS balance | after 2 + 4 weeks
  kind, frequency, duration, outcome of ADR
Change of 13 common symptoms of nervous restlessness | after 2 + 4 weeks
  Questionnaire on 13 common symptoms of nervous restlessness in children
Change of the impact of the child´s complaints on daily family life (VAS) | after 2 + 4 weeks
  Visual Analogue Scale (VAS)to assess the impact of the child´s complaints on daily family life

CONTACTS AND LOCATIONS:
Overall Officials: Anja Braschoss, MD, Study Director — Pascoe Pharmazeutische Praeparate GmbH
Locations (1):
- multiple German Paediatric Practices, Giessen, Hesse, Germany